CLINICAL TRIAL: NCT02420418
Title: The Effect of N- Acetylcysteine on Inflammatory and Oxidative Stress Biomarkers in Patients With Tobacco Use Disorders and Bipolar Disorders ..
Brief Title: The Effect of N- Acetylcysteine on Inflammatory and Oxidative Stress Biomarkers
Acronym: nac
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Sandra Odebrecht Vargas Nunes, PHD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ULondrina
Record Dates: First submitted 2015-01-22; First posted 2015-04-17 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Bipolar Disorder
Keywords: Tobacco use disorder and bipolar disorders; N-acetylcysteine; Oxidative stress; inflammation
MeSH Terms: conditions — Bipolar Disorder; Tobacco Use Disorder; Inflammation | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAC ( baseline )and 12 week (Active Comparator): subjects with tobacco use disorder (TUD) and bipolar disorders who will receive N-acetyl-cysteine (NAC) or placebo at baseline for a period of 12 weeks The participants with TUD (n=72) and they will receive a 1800mg per day of NAC or matching placebo .
  There will be asses laboratory examinations for inflammatory and oxidative stress biomarkers at baseline and at 12 week
  Interventions: Dietary Supplement: N-acetyl-cysteine (NAC)
- placebo ( baseline ) and 12 week (Placebo Comparator): subjects with tobacco use disorders (TUD and bipolar disorders who will receive N-acetyl-cysteine (NAC) or placebo for a period of 12 weeks.
  The participants with TUD and bipolar disorders (n=72) and they will receive a 1800mg per day of NAC or matching placebo .
  There will be assessed laboratory examinations for inflammatory and oxidative stress biomarkers at baseline and at 12 week
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: N-acetyl-cysteine (NAC) — Patients will be randomly allocated into two groups, double-blind, to receive NAC or placebo for a period of 12 weeks. All groups remain receiving maintenance treatment in outpatient smokiing cessation. The dosage will be fixed 1800 mg/day of NAC administered in capsules taken 2 before breakfast and 2 before dinner is equal doses.
  Arms: NAC ( baseline )and 12 week
Other: Placebo — Patients will be randomly allocated into two groups, double-blind, to receive NAC or placebo for a period of 12 weeks. All groups remain receiving maintenance treatment in smoking cessation service
  Arms: placebo ( baseline ) and 12 week

SUMMARY:
Background: . Bipolar disorders and tobacco use disorder are top of the causes of disability and mortality worldwide Objective: The aim of this study was to evaluate N-acetyl-cysteine (NAC) as an adjunctive treatment in patients with bipolar .disorders and tobacco use disorder (TUD)

, to determine whether NAC reduces alterations in biomarkers of inflammatory and oxidative stress Methods: This study will be conducted as a double-blind, randomized, placebo controlles add NAC or placebo for .bipolar disorders and tobacco use disorder at Londrina State University, Brazil.

DETAILED DESCRIPTION:
Tobacco use disorder and bipolar disorders are top of the causes of disability and mortality worldwide. The aim of this study was to evaluate N-acetyl-cysteine (NAC) as an adjunctive treatment in patients with Tobacco use disorder with comorbid bipolar disorder ( (N=72 NAC/placebo ) recruited from outpatients smoking cessation unit at Londrina State University, Brazil.

The design was a randomized, double-blind, placebo controlled clinical trial of 12 weeks of adjunctive treatment with N-acetyl-cysteine (NAC), 1800mg/day. Participants will be patients with bipolar disorders with and without TUD, they will allocated to one of two groups at random to receive NAC or placebo For the evaluation of oxidative stress biomarkers will be assess among others malondialdehyde (MDA), lipid hydroperoxide,nitric oxide metabolites (NOx), antioxidant potential total plasma (TRAP), advanced oxidation protein products (AOPP), superoxide dismutase (SOD), catalase, the total glutathione (GSH) and oxidized (GSSG), paraoxonase (PON 1) activity thiol group (SH-group).For the evaluation of inflammation biomarkers will be analyze : BDNF, GM-CSF, IFN-γ, IL-1β, IL-10, IL-12 (p70), IL-13, IL-15, IL-17, IL-1RA, IL-2, IL-2R, IL-4, IL-5, IL-6,IL-6R, IL-7, IL-8, Leptin, TNF-α, TNF-RI, TNF-RII, high-sensitivity C-reactive protein (hs-CRP), erythrocytes sedimentation rate (ESR), homocysteine, haptoglobin, albumin , uric acid and fibrinogen.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study participants must be motivated smokers to stop tobacco use
* Age greater than or equal to 18 and less than 65 years
* Both sexes
* All races
* Capacity to consent to the study and carefully follow the guidelines and procedures and sign the term of free and informed consent .
* Will be included with comorbid bipolar, depressive and anxiety disorder with tobacco use by more than 20 cigarettes per day, and a control group without these mood disorders and without tobacco use disorder.

Exclusion Criteria:

* We excluded any subjects with: abnormal blood values on the following laboratory tests: *hemogram, aspartate transaminase (AST), alanine transaminase (ALT), urea and creatinine

  * other actual and life-time axis-I diagnoses (including schizophrenia, psycho-organic syndromes, delirium, dementia, amnestic, and other cognitive disorders)
  * medical illness, including HIV and hepatitis B and C, (auto)immune disorders
  * immune modulatory drugs, e.g. glucocorticoids and use of antioxidants.
* These situations can affect an inflammatory and / or immune process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The effect of N- acetylcysteine on oxidative stress biomarkers in patients with tobacco use disorders and bipolar disorders | 12 weeks
  The design was a randomized, double-blind, placebo controlled clinical trial of 12 weeks of adjunctive treatment with N-acetyl-cysteine (NAC). For the evaluation of oxidative stress biomarkers will be assess among others malondialdehyde (MDA), lipid hydroperoxide,nitric oxide metabolites (NOx), antioxidant potential total plasma (TRAP), advanced oxidation protein products (AOPP), superoxide dismutase (SOD), catalase, the total glutathione (GSH) and oxidized (GSSG), paraoxonase (PON 1) activity thiol group (SH-group).
The effect of N- acetylcysteine on inflammatory in patients with tobacco use disorders and bipolar disorders | 12 weeks
  For the evaluation of inflammation biomarkers will be analyze : BDNF, GM-CSF, IFN-γ, IL-1β, IL-10, IL-12 (p70), IL-13, IL-15, IL-17, IL-1RA, IL-2, IL-2R, IL-4, IL-5, IL-6,IL-6R, IL-7, IL-8, Leptin, TNF-α, TNF-RI, TNF-RII, high-sensitivity C-reactive protein (hs-CRP), erythrocytes sedimentation rate (ESR), homocysteine, haptoglobin, albumin , uric acid and fibrinogen.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Landucci Bonifácio, MS, Principal Investigator — Universidade Estadual de Londrina; Ana Carolina Rossaneis, PhD, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- State University of Londrina, Londrina, Paraná, Brazil

REFERENCES:
- [Derived] Machado RCBR, Vargas HO, Baracat MM, Urbano MR, Verri WA Jr, Porcu M, Nunes SOV. N-acetylcysteine as an adjunctive treatment for smoking cessation: a randomized clinical trial. Braz J Psychiatry. 2020 Sep-Oct;42(5):519-526. doi: 10.1590/1516-4446-2019-0753. PMID 32725102